CLINICAL TRIAL: NCT00196170
Title: Multicenter Prospective Randomized Clinical Study Comparing Radiofrequency- vs. Cryo-Ablation in Typical Isthmus-Dependent Atrial Flutter
Brief Title: Randomized Study of Radiofrequency- vs. Cryo-Ablation for Typical Isthmus-Dependent Atrial Flutter
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. C00303
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-03

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 8mm tip ablation catheter for ablation of cavotricuspid isthmus
  Interventions: Procedure: RF ablation of the cavo-tricuspid isthmus
- 2 (Experimental): irrigated tip ablation catheter for ablation of cavotricuspid isthmus
  Interventions: Procedure: irrigated tip radiofrequency ablation of the cavo-tricuspid isthmus
- 3 (Experimental): cryo 10mm tip ablation catheter for ablation of cavotricuspid isthmus
  Interventions: Procedure: cryo ablation of the cavo-tricuspid isthmus
- 4 (Experimental): Cryo 6.5mm tip ablation catheter for ablation of cavotricuspid isthmus
  Interventions: Procedure: cryo 6.5mm tip ablation of the cavotricuspid isthmus

INTERVENTIONS:
Procedure: RF ablation of the cavo-tricuspid isthmus — 8mm tip ablation catheter is used for the radiofrequency ablation of the cavo-tricuspid isthmus in typical atrial flutter
  Arms: 1
Procedure: cryo ablation of the cavo-tricuspid isthmus — Cryo 10mm tip ablation catheter is used for the cryo ablation of the cavo-tricuspid isthmus in typical atrial flutter
  Arms: 3
Procedure: irrigated tip radiofrequency ablation of the cavo-tricuspid isthmus — irrigated tip ablation catheter is used for the radiofrequency ablation of the cavo-tricuspid isthmus in typical atrial flutter
  Arms: 2
Procedure: cryo 6.5mm tip ablation of the cavotricuspid isthmus — cryo 6.5mm tip ablation catheter is used for the cryo ablation of the cavo-tricuspid isthmus in typical atrial flutter
  Arms: 4

SUMMARY:
This randomized study compares two energy sources for the catheter based ablation of typical isthmus-dependent atrial flutter: The (standard) radiofrequency (RF) ablation technique and the cryo-ablation technique regarding the acute and long term efficacy and safety.

DETAILED DESCRIPTION:
This randomized study compares two energy sources for the catheter based ablation of typical isthmus-dependent atrial flutter: The (standard) radiofrequency (RF) ablation technique and the cryo-ablation technique. The RF ablation of typical atrial flutter has become a standard approach with very high curing rates and low complication incidence. However, ablation with RF is painful since the underlying cardiac tissue heats up (up to 70-80°C inside the tissue) and especially the target of ablation in typical atrial flutter, the so-called cavo-tricuspid isthmus, is a very pain-receptive area. Cryo-ablation, which destroys tissue by freezing it down to -80 to -90°C, is thought to be less painful or even painless with the same efficacy than RF ablation.

The acute and long term (6 months follow-up, non-invasive) efficacy and safety is the combined endpoint.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* documented atrial flutter which is most probably typical isthmus dependent atrial flutter
* informed written consent

Exclusion Criteria:

* prior ablation for atrial flutter
* concomitant arrhythmia which is treated during the same ablation procedure
* prior MAZE operation
* contra indication for catheterization
* physical or psychiatric disorder making participation in the study impossible
* pregnancy
* prior participation in the study
* participation in another study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2003-05; Primary Completion 2008-04 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Acute Efficacy (bidirectional cavotricuspid isthmus block) | bidirectional cavotricuspid isthmus block
Long-term efficacy (6 months FU freedom of typical atrial flutter) | 6 months
Mortality | 6 months

SECONDARY OUTCOMES:
Patients' pain scores during ablation | while hospitalisation
Safety of ablational devices | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Claus Schmitt, MD, Study Chair — Deutsches Herzzentrum Muenchen; Bernhard Zrenner, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (4):
- Germany (4):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Deutsches Herzzentrum Muenchen, Munich
  - Westfälische Wilhelms-Universitaet Muenster, Münster
  - Klinikum Nuernberg Sued, Nuremberg